CLINICAL TRIAL: NCT04598646
Title: The Harmonized Interventions to Maintain Health Via Appropriate Risk Factor Modification and Lifestyle Changes in Pediatric, Adolescent and Young Adult Cancer Survivors Pilot Study
Acronym: HIMALAYAS-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-5391.0
Record Dates: First submitted 2020-08-27; First posted 2020-10-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Cardiotoxicity; Cancer
Keywords: Adolescents and Young Adults; Exercise Therapy; Behavioral and Peer Support; Cardiac Rehabilitation; Cancer Survivor
MeSH Terms: conditions — Heart Failure; Cardiotoxicity; Neoplasms; Behavior | interventions — Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cario-Oncology Rehabilitation (CORE) (Experimental): CORE consists of exercise therapy, CVD risk factor management, and behavioural support for 3 months.
  Exercise therapy: Staff will prescribe and deliver a standardized, yet individually tailored (based on CPET results), aerobic exercise programs consisting of two days of supervised, facility- and home-based high-intensity interval training (HIIT) and one day of supervised home-based moderate-intensity continuous training (MICT) per week. Exercise HRs and durations will be monitored using an accurate commercially available wrist-worn HR monitor and PA tracker.
  CVD risk factor management: CVD risk factors will be assessed and treated according to Canadian guidelines.
  Behavioural support: All participants will receive a planned sequence of educational and instructional material via email and ongoing PAYA-CS tailored education and peer support during the follow-up period using a peer support online system.
  Interventions: Behavioral: Cardio-oncology Rehabilitation (CORE)
- Support (Experimental): The Support group will receive the behavioural support only. The timing and nature of all education, information provided to Support participants will be identical to what is provided to CORE participants. All Support participants will receive the same wrist-worn HR monitor and PA tracker as the CORE participants and will be given the challenge of meeting and maintaining the updated PA guidelines for cancer survivors (i.e., 90 to 150 minutes of moderate to vigorous intensity PA per week).
  Interventions: Behavioral: Support

INTERVENTIONS:
Behavioral: Cardio-oncology Rehabilitation (CORE) — Exercise therapy, CVD risk factor management for the first 6 months (as per current standards in CR models) and behavioural support for the entire 2-year intervention period
  Arms: Cario-Oncology Rehabilitation (CORE)
Behavioral: Support — Behavioural support via professionals and peer support and recommended physical activity guidelines for cancer survivors, to encourage physical activity.
  Arms: Support

SUMMARY:
Cardiovascular disease (CVD) is a major contributor to morbidity and mortality in pediatric, adolescent and young adult (AYA) cancer survivors (hereafter referred to as PAYA-CS). Exercise is a cornerstone of CVD prevention and treatment; yet, exercise has not been adopted as a standard of care in PAYA-CS at high CVD risk. The HIMALAYAS trial is designed to evaluate the feasibility and preliminary impact of an exercise-based CR on cardiovascular (CV) and psychosocial health, as well as CVD risk, in PAYA-CS with mild heart dysfunction (stage B heart failure (SBHF)). The primary objective of the HIMALAYAS pilot study is to assess the feasibility of a two-phase randomized controlled trial designed to evaluate impact of a 'CR-like' cardio-oncology rehabilitation (CORE) intervention on CV, psychosocial, and behavioural outcomes at 6 and 24 months, compared to behavioural support only (Support) in PAYA-CS. Screened PAYA-CS without SBHF and those with SBHF who do not participate in the RCT will be enrolled in a passive behavioural support (Support) group. The primary outcome is study feasibility, defined according to three primary criteria (i.e., participant recruitment, safety, and adherence). Secondary outcomes include additional feasibility metrics (e.g., intervention safety and tolerability) and exploratory efficacy outcomes including peak cardiorespiratory fitness (VO2peak), cardiac function (e.g., global longitudinal strain (GLS)), CVD risk factor control (e.g. insulin resistance), and patient-reported outcomes (e.g. anxiety). Our central hypothesis is that the conduct of a larger RCT comparing the impact of CORE versus non-intervention control will be feasible indicated by the achievement of our primary feasibility criteria. Our exploratory hypothesis is that we will generate preliminary evidence that CORE can improve VO2peak, cardiac function, CVD risk factor, and patient-reported outcomes over 6- and 24-month timepoints, relative to control.

DETAILED DESCRIPTION:
Over 90,000 North Americans are diagnosed with cancer before the age of 40. Improved cancer therapies have led to an exponential growth in the number of pediatric, adolescent, and young adult cancer survivors (PAYA-CS) who are expected to live 50-60 years beyond diagnosis. However, PAYA-CS are at increased risk of developing multiple cancer- and treatment-related morbidities including poor fitness (e.g., low VO2peak), hypertension (HTN), diabetes, and poor mental health, which all contribute to premature cardiovascular disease (CVD). The prevalence of CVD events (e.g. heart failure, heart attack, stroke) is up to 23.8% in adult survivors of pediatric cancers with long term follow-up after treatment. The incidence of subclinical CVD, which is a precursor to CVD events, is even higher in PAYA-CS; up to 40%, 11%, and 5% experience subclinical cardiomyopathy measured by abnormal global longitudinal strain (GLS), diastolic dysfunction (DD) or mild reduction in left ventricular ejection fraction (LVEF), respectively, and 18% experience reduced aerobic fitness. The treatment of modifiable CVD risk factors must be considered a fundamental target for improving CVD health-related outcomes in PAYA-CS. To this end, exercise and best-practices for CVD risk factor modification are integral to a cardiac rehabilitation (CR) model. Traditional cardiac rehabilitation models for patients with CVD (consisting of exercise, CVD risk factor treatment, and patient education) are safe and effective in improving HRQoL, morbidity, and mortality risk. However, by virtue of their age and low short-term CVD risk, PAYA-CS do not meet traditional criteria for initiating CR and are less likely to receive treatments to reduce CVD risk.

PAYA-CS with stage B heart failure (SB¬HF): (1) are at high risk for subsequent HF/CVD death; (2) have lower cardiopulmonary fitness; and (3) are more likely to benefit from CVD risk factor management. Considering that PAYA-CS have an estimated 33% prevalence of SBHF, this vulnerable cohort of cancer survivors represent an opportunity for intervention that is highly feasible and potentially impactful. Exercise is a preferred method for optimizing health and survival in PAYA-CS. However, we need models that safely and effectively deliver exercise interventions that meet the unique needs of this population. The cardio-oncology rehabilitation (CORE) model is an intervention that would provide PAYA-CS with SBHF a supervised and home-based exercise therapy, CVD risk factor modification, and behavioural support to reduce the risk of CVD. Nevertheless, due to the ambitious nature of the study, it is vital that we conduct a pilot version of the study to determine the feasibility and needed changes to achieve the best possible results.

The primary objective of the HIMALAYAS pilot study is to assess the feasibility, safety, and tolerability of a (1) two-arm RCT-based comparison of the CORE and Support interventions in PAYA-CS with SBHF, and (2) parallel passive behavioural support (PBS) cohort of PAYA-CS at high-risk of cancer-related CVD. The exploratory objectives of the study include (1) to compare the changes in primary exploratory outcome (VO2peak) and secondary exploratory outcomes (markers of cardiac function, CVD risk factor management, and patient-reported outcomes) between a CORE and Support intervention for PAYA-CS from baseline (T0) to 6-month (T1) follow-up and (2) to compare the changes in the primary and secondary exploratory outcomes between (1) CORE and Support from T0 to 12-month (T2) and 24-month (T3) follow-up, and (2) CORE, Support, and PBS from T0 to T3.

Cardio-oncology Rehabilitation (CORE) Group: CORE consists of exercise therapy, CVD risk factor management for the first 6 months (as per current standards in CR models) and behavioural support for the entire 2-year intervention period.

Support Group: The Support group will receive the behavioural support only. The timing and nature of all education, information, and peer support provided to Support participants will be identical to what is provided to CORE participants. The key difference in the long-term behavioural support strategy between CORE and Support participants is how weekly exercise goals are defined. Unlike the CORE participants who will be encouraged to use the personal activity intelligence (PAI) Score, Support participants will be given the challenge of meeting and maintaining the updated physical activity (PA) guidelines for cancer survivors (i.e., 90 to 150 minutes of moderate to vigorous-intensity PA per week).

Passive Behavioural Support (PBS) Groups: All PBS cohort participants will receive the same wrist-worn heart rate monitor and PA tracker as the CORE and Support participants. However, PBS participants will be blindly randomized to one of two passive behavioural support interventions (PBS1 and PBS2). PBS1 participants will be asked to download the same PAI Health application as CORE participants and will similarly be given the challenge of meeting and maintaining a weekly PAI Score ≥100 throughout the 18-month follow-up period. PBS2 participants will be asked to download and use the Map My Walk (Under Armour, Baltimore) application and will be challenged to meet and maintain the updated PA guidelines for cancer survivors (i.e., 90 to 150 minutes of moderate to vigorous intensity PA per week).

ELIGIBILITY:
Inclusion Criteria:

* Be a PAYA-CS, defined as ≤39 years of age at the time of cancer diagnosis;
* Be 18-45 years of age at the time of enrolment;
* Received cancer treatment(s) with known cardiovascular risks (e.g. anthracyclines, radiotherapy, trastuzumab, platinum-based agents, vascular endothelial growth factor inhibitors, tyrosine kinase inhibitors);
* Be cancer-free at the time of enrollment.
* Diagnosed with SBHF prior to or at baseline (LVEF<53/54%, GLS >-18%, or diastolic dysfunction).

Exclusion Criteria:

* An absolute or relative contraindication to exercise according to the American College of Sports Medicine (ACSM) guidelines;
* Untreated physical or mental health concerns that preclude safe and effective exercise participation;
* Established CVD (excluding mildly reduced LVEF as described above);
* Be currently engaging in high-intensity exercise (>1 high-intensity exercise session per week);
* Substantial barriers to completing study protocol (e.g. living too far away and being unable to attend testing and exercise training sessions) or unwillingness to comply with the study protocol (e.g. individual intends to start performing regular HIIT exercise regardless of randomization).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Patient Access and Recruitment (feasibility target: >50% of eligible participants) | Throughout study recruitment, up to 2 years
  Defined as the percent of consenting patients based on the total number of otherwise eligible participants (OEP; patients meeting all eligibility criteria) approached
Testing- and intervention-related serious adverse events (feasibility target: none) | Initiation through end of study recruitment 12 months
  Defined as the number and frequency of testing- and intervention-related serious adverse events (SAEs) according to the Common Terminology Criteria for Adverse Events
Patient exercise adherence (feasibility target: >=70% of prescribed) | Initiation throughout end of CORE intervention at a maximum of 6 months post-randomization
  Defined as relative dose intensity as the percent of total dose of exercise performed relative to the total planned dose prescribed and quantified according to metabolic equivalents

SECONDARY OUTCOMES:
Patient identification rate (feasibility target: >=50% of OEP) | Initiation through end of study recruitment 12 months
  Defined as the average number of OEP identified each month
Baseline assessment rate (feasibility target >=90% of consenting participants) | Initiation through end of study recruitment 12 months
  Defined as the percent of consenting patients who successfully complete baseline assessments based on the total number of consenting patients
Testing- and intervention-related non-serious adverse events (feasibility target <=20% of consenting participants) | Initiation through end of study recruitment 12 months
  Defined as the number and frequency of testing- and intervention-related non-serious adverse events
Testing performance (feasibility target >=95% of consenting participants) | Initiation through end of study recruitment 12 months
  Defined as the percent completion of all cardiopulmonary exercise tests (CPETs) tests at baseline (T0) and primary follow-up (T1)
Testing modality adaptation (descriptive) | Initiation throughout end of CORE intervention at a maximum of 6 months post-randomization
  Defined as the percent of all tests which are adapted for functional or safety reasons
Training modality adaptation (descriptive) | Initiation throughout end of CORE intervention at a maximum of 6 months post-randomization
  Defined as the percent of all exercise sessions which are adapted for functional or safety reasons
Permanent treatment discontinuation (feasibility target <=15% of participants) | Initiation throughout end of CORE intervention at a maximum of 6 months post-randomization
  Defined as the percent of patients who discontinue intervention participation prior to the planned end of the intervention period
Treatment interruption (feasibility target <=15% of participants) | Initiation throughout end of CORE intervention at a maximum of 6 months post-randomization
  Defined as the percent of patients who miss =>3 consecutive sessions within the intervention period
Dose modification (feasibility target <=25% of participants) | Initiation throughout end of CORE intervention at a maximum of 6 months post-randomization
  Defined as the percent of exercise sessions requiring a dose reduction during training (i.e., intensity or duration) relative to the total number of sessions completed. Total number of exercise sessions with a reduction in intensity or a reduction in duration will be combined into the numerator when calculating the percentage of affected sessions.
Early session termination (feasibility target <=25% of participants) | Initiation throughout end of CORE intervention at a maximum of 6 months post-randomization
  Defined as the percent of exercise sessions requiring unplanned early termination
Pretreatment intensity modification (feasibility target <=25% of participants) | Initiation throughout end of CORE intervention, an average of 6 months
  Defined as the percent of sessions which required pre-exercise modification of the target exercise intensity due to a pre-exercise screening indication (e.g., fatigue, pain)
Exercise compliance (feasibility target >=70% of prescribed) | Initiation throughout end of CORE intervention at a maximum of 6 months post-randomization
  Defined as the percent of exercise sessions completed based on the total number of sessions prescribed.
Medication compliance (feasibility target >=70% of prescribed) | Initiation throughout end of CORE intervention at a maximum of 6 months post-randomization
  Defined as the percent of pharmaceutical doses taken based on the total number of doses prescribed (applicable only to those that are provided pharmaceutical therapy for CVD risk factor modification.
Behavioural compliance (feasibility target >=70% of prescribed) | Initiation throughout end of study, an average of 2 years
  Defined as the percent of behavioural support resources accessed, based on the number of doses prescribed
Physical activity compliance (feasibility target >=70% of prescribed) | Initiation throughout end of study, an average of 2 years
  defined as the average number of participants achieving their weekly PA goals of meeting and maintaining either a PAI-Score of ≥100 or weekly cancer exercise guidelines (i.e., 90 to 150 minutes of moderate to vigorous intensity PA per week).
Attrition (feasibility target <=15% loss to follow-up) | Initiation throughout end of 6 months post-intervention period
  Defined as the percent loss to follow-up (not completing follow-up assessments)

OTHER OUTCOMES:
VO2peak | baseline, 6-, 12- and 24-month follow ups
  VO2peak measured by CPET
Cardiac function | baseline, 6-, 12- and 24-month follow ups
  2D LVEF measured by echocardiogram
Cardiac function | baseline, 6-, 12- and 24-month follow ups
  3D LVEF measured by echocardiogram
Cardiac function | baseline, 6-, 12- and 24-month follow ups
  GLS measured by echocardiogram
Resting blood pressure | baseline, 6-, 12- and 24-month follow ups
  Measured with an average of 3 readings (after discarding an initial test reading) by an automated measurement device as per the Hypertension Canada guidelines.
Resting heart rate | baseline, 6-, 12- and 24-month follow ups
  Measured with an average of 2 readings taken via ECG during the resting period during the cardiac screening procedures.
Hyperlipidemia | baseline, 6-, 12- and 24-month follow ups
  Measured through fasting cholesterol profile and Apo B levels
Diabetes and diabetes risk | baseline, 6-, 12- and 24-month follow ups
  Measured through fasting glucose
Diabetes and diabetes risk | baseline, 6-, 12- and 24-month follow ups
  Measured through whole-body insulin sensitivity (Matsuda index)
Diabetes and diabetes risk | baseline, 6-, 12- and 24-month follow ups
  Measured through hepatic insulin sensitivity (HOMA-IR)
Diabetes and diabetes risk | baseline, 6-, 12- and 24-month follow ups
  Measured through pancreatic beta-cell function (ISSI-2).
Diabetes and diabetes risk | baseline, 6-, 12- and 24-month follow ups
  Measured through fasting insulin
Physical activity | baseline, 6-, 12- and 24-month follow ups
  Measured through Godin Leisure Time PA Questionnaire (GLTPAQ). Score of >24 = active, score of 14-23 = moderately active, score of <14 = insufficiently active
Physical activity | baseline, 6-, 12- and 24-month follow ups
  Measured through wrist-worn heart rate with physical activity monitor
Social support | baseline, 6-, 12- and 24-month follow ups
  Measured using the Social Support Survey-Clinical (SSS-C) form, a 5-item survey designed to measure five dimensions of social support (listening, task challenge, emotional reality confirmation, and tangible assistance); higher score = more social support
Exercise self-efficacy | baseline, 6-, 12- and 24-month follow ups
  Measured using the Multidimensional Self-Efficacy for Exercise Scale (MSES) to measure three behavioural subdomains: task, scheduling, and coping; Scale 0-90, higher score indicates higher self-efficacy for exercise.
Dietary habits | baseline, 6-, 12- and 24-month follow ups
  Measured using the National Health and Nutrition Examination Survey (NHANES) Food Frequency Questionnaire (FFQ), a 139-item, semi-quantitative inventory to assess the potential influence of dietary changes on primary and secondary outcomes.
Smoking status | baseline, 6-, 12- and 24-month follow ups
  Measured using self-reported measures to determine the potential influence of changes in smoking habits on primary and secondary outcomes.
Anxiety | baseline, 6-, 12- and 24-month follow ups
  Measured using the Generalized Anxiety Disorder (GAD-7), a 7-item inventory that assesses 2-week anxiety symptom frequency on a 0-3 scale, with higher scores reflecting higher symptom frequency. A cut-off of ≥10 indicates some degree of clinical anxiety
Depression | baseline, 6-, 12- and 24-month follow ups
  Measured using the Patient Health Questionnaire (PHQ-9), a 9-item inventory that assesses 2-week depressive symptom frequency on a 0-3 scale, with higher scores reflecting higher symptom frequency. The PHQ-9 has been validated in cancer survivors using a cut-off of ≥8 to indicate some degree of clinical depression.
Health-related quality of life | baseline, 6-, 12- and 24-month follow ups
  Measured using the Medical Outcomes Survey Short-Form, (SF-12).
Therapeutic alliance | baseline, 6-, 12- and 24-month follow ups
  Measured using the Working Alliance Inventory Short-Revised (WAI-SR) form. Increased score indicates therapeutic alliance.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada